CLINICAL TRIAL: NCT05778669
Title: Early Childhood Intervention to Reduce Deficits of Underprivileged Children - Follow-up Study
Brief Title: KeySteps@JC Phase One Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: KeySteps@JC 1.0 FU
Record Dates: First submitted 2023-02-19; First posted 2023-03-21 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Child Development
Keywords: Community child health; Child development; Motor performance; Nutrition; Physical activity; Sleep; KeySteps; Long term benefits; Sustainable effects
MeSH Terms: conditions — Motor Activity | interventions — Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort Group: Longitudinal follow-up intervention: Monitoring of medical, health and psychosocial conditions through questionnaires, on-site assessments and medical record checking.
  Interventions: Other: Monitoring of medical, health and psychosocial conditions

INTERVENTIONS:
Other: Monitoring of medical, health and psychosocial conditions — Questionnaires will be used to collect information including children's health and psychosocial conditions, academic performance, and family demographics.
  On-site assessments including general health and learning assessments.
  Tracking of medical and health-related events of participants will be performed through the existing health care system.

SUMMARY:
This proposed study is a 5-year follow-up study of "KeySteps Phase One Study", which focused on bridging the gap between students from privileged and underprivileged families.

This study will investigate the long-term effects of early childhood interventions provided during the kindergarten stage on primary school children and their families and track the health conditions and development of the Project children in their primary school stage.

Cohort students of "KeySteps Phase One Study" will be invited to join this follow-up study. Data including children's health and psychosocial conditions, academic performance, and family demographics will be collected. In addition, subjects will receive on-site assessments on general health and learning. Medical and health-related events of subjects will be tracked through the existing health care system.

DETAILED DESCRIPTION:
Emerging evidence suggests that childhood is a sensitive period during which socioeconomic conditions become biologically embedded despite current circumstances during adulthood. Children with socioeconomic disadvantages are vulnerable to numerous health problems later in life, including cardiovascular and respiratory diseases. In both children and adults, the associations between socioeconomic status (SES) and life outcomes are monotonic or graded, such that individuals higher in the socioeconomic hierarchy enjoy better health status and well-being than those individuals one level below.

Socioeconomic disparities in developmental trajectories can be observed in the early years of life and this has necessitated a closer look at the childhood family environment. Families who are confronting socioeconomic struggles also tend to have higher levels of conflict, harsh restrictive parenting styles, chaotic or neglectful parenting, as well as inadequate emotional nurturing. Children reared in family environments marked by these adverse social conditions also tend to show elevated physiological responses to stress.

Continued urban development in Hong Kong has led to a simultaneous increase in economic indices, but also widen the socioeconomic gaps between social groups. Parallel to epidemiological patterns in other countries, the Child Health Survey documented that children from low SES families in Hong Kong were also more likely to suffer from worse physical and psychological health. Early sleep deprivation and overuse of digital devices were also more prevalent among the lower social class which resulted in problematic behaviour and learning.

The original project ("KS Phase One Study") focused on bridging the gap between students from privileged and underprivileged families. Results showed that there were improvements in school readiness and holistic development of children of the underprivileged children during their kindergarten stage. The promising findings worth further follow up to study the long-term benefits and sustainable effects, if any, in different dimensions of child development in longer term. The proposed follow-up study will recruit those subjects who had joined the original study "KS Phase One Study" as main cohort in the 32 Project schools in Sham Shui Po and Tin Shui Wai previously. Most families in those areas were with lower SES.

The hypothesis of the study is early interventions to children, families and schools during the kindergarten stage will have positive effects on shaping the trajectories in children and their families during the primary school stage. Questionnaires will be used collect information including children's health and psychosocial conditions, academic performance, and family demographics. Children general physical health and learning assessments will be carried out on-site. Their medical and health-related events will be tracked through the existing health care system.

Since all assessments used in this study are non-invasive, there should be no foreseeable major safety concern to the study subjects. Should there be unanticipated problems involving risk to study subjects or others or severe adverse events, they will be reported to the Research Ethics Committee responsible for overseeing this study (Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster) according to the set guidelines.

The analysis plan will be guided by the research aims and the hypothesis. Categorical data will be summarised with counts (percentages), continuous data with normal distribution will be summarised with mean (standard deviation [SD]) and median (interquartile or entire range) will be reported for other continuous data. Independent variables will be screened for statistically significance with the outcomes measured prior to conducting multilevel and multivariate regression analyses.

The Principal Investigator is responsible for ensuring data obtained from this research is accurate, complete and reliable. All information and data collected throughout the course of this study will remain strictly confidential to the research team members and will be used solely for research purposes. Identifiable information (e.g. names and identity card numbers) will be kept confidential and data collected in this study will be password-protected and restricted to designated research personnel. Personal records, to the extent of the applicable laws and regulations, will not be made publicly available. In the event of any report, presentation and/or publication of findings regarding this study, subjects' identity will not be disclosed. This study will be conducted in compliance with the protocol, Declaration of Helsinki and other applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Children and their families of the KS Phase One Study cohort in Academic Year 2018-19
* Children and their families are willing to join this follow-up study

Exclusion Criteria:

* Children and their families withdrew themselves from KS Phase One Study (KeySteps@JC - Early Child Intervention (KSJC) previously
* Children cannot understand Chinese
* Children's parents cannot understand Chinese
* Children who are not studying primary schools in Hong Kong

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All cohort subjects of "KeySteps Phase One Study" [KeySteps@JC - Early Child Intervention (KSJC)] will be invited for this follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 1486 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Growth and development of the children | 5 years
  Children's body height, weight, blood pressure, body fat and physical performance (cardiorespiratory endurance, muscle strength and endurance, flexibility according to the Hong Kong Education Bureau School Physical Fitness Award Scheme guidelines).
Nutritional status of the children | 5 years
  Assessing the nutritional status and dietary habits with the food frequency questionnaire (electronic version)
Activity and sleep condition of the children | 5 years
  Assessing the physical activity level and sleep duration with the activity monitoring device (Actigraph)
Psychosocial development of the children | 5 years
  Different scales will be used to assess the child's psychosocial development namely the Strength and Difficulties Questionnaire (SDQ), Paediatric Quality of Life (PQoL), Chinese Strengths and Weaknesses of Attention Deficit Hyperactivity Disorder Symptoms and Normal Behaviour Scale (SWAN).

SECONDARY OUTCOMES:
Parent Well-Being and Coping | 5 years
  The Parental Stress Scale (PSS) and questions on perceived financial strain will be used to assess the stress level of parents.
Family Functioning | 5 years
  The Chinese Parent-Child Conflicts Tactic Scale (CTSPC) and questions related to parental involvement in children's education will be used to assess family functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick IP, MBBS, MPH, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No